CLINICAL TRIAL: NCT05738421
Title: THE IMPACT OF TRACHEAL TUBE ON SWALLOWING IN POST-OPERATIVE HEAD AND NECK CANCER PATIENTS: SCINTIGRAPHIC ANALYSIS
Brief Title: Tracheal Tube and Swallowing After Head and Neck Surgery
Status: Recruiting | Type: Observational
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Responsible Party: Principal Investigator, Galli Jacopo, Full Professor, Director of Otorhinolaryngology Unit, Fondazione Policlinico Universitario Agostino Gemelli IRCCS
Other Study IDs: 4459
Record Dates: First submitted 2023-02-01; First posted 2023-02-22 (Actual); Last update posted 2024-10-04 (Actual); Status verified 2024-10

CONDITIONS: Dysphagia
MeSH Terms: conditions — Deglutition Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: fiberoptic endoscopic evaluation of swallowing — Questionnaire, FEES, OPES

SUMMARY:
The present study was designed as a cross-sectional observational study providing the enrollment of tracheostomized patients undergoing major oncological surgery for head-neck cancer.

Aims:

* to provide objective data on the bolus transit during swallowing in tracheostomized patients with tracheal tube and without tracheal tube closing directly the tracheal stoma with a plaster, in order to sustain the choice to preserve the TT in dysphagic patients after oncologic surgery for more security during swallowing rehabilitation or adjuvant treatment.
* to evaluate the features of swallowing, specifically bolus transit, in patients affected by head and neck cancer who underwent major oncological surgery.

DETAILED DESCRIPTION:
In the last twenty years, a wide and conflicting literature discussed about the impact of the presence of a tracheal tube (TT), even if occluded, on the swallowing function. Early the majority of authors agreed to target the tracheal tube as the cause of aspiration basing on several mechanisms, first of all the decrease of laryngeal elevation. Nevertheless over time, new researches had open to different results. In 2010 Leder et al. [1] demonstrated the absence of a causal relationship between tracheotomy and aspiration status in 25 patients who underwent fiberoptic endoscopic evaluation of swallowing (FEES) and more recently Kang et al. [2] showed by Videofluoroscopic Swallow Study (VFSS) that the swallowing parameters related to laryngeal elevation, pharyngeal constriction, and esophageal opening did not changed significantly between patients with and without tracheostomy. However until now the study samples and methods employed to analyze the same purpose were heterogenous. At first the earlier researches were mostly conducted immediately after tracheostomy, while the latest ones on cases with stabilized tracheal stoma [3]. Furthermore, the possible mechanisms hypothesized to explain the increased risk of aspiration were the same both for the studies about the effect of TT occlusion status and the ones about the presence of TT. Dysphagia is a dysfunction that deeply impacts especially the patient's post-surgery recovery, particularly dysphagia is the most common short-term and long-term sequela in subjects undergoing head and neck oncologic surgery. On this regard the tracheostomy and tracheal tube represent an unquestionably security condition and a security device respectively. At a time when the hospitalization is getting shorter and the swallowing rehabilitation training is mainly carried out in the outpatient setting, it is even more important to clarify the real impact of tracheal tube. Anyhow, to date the often-held assumption that tracheotomy and placement of an occluded tracheotomy tube, by themselves, increase incidence of aspiration was not supported by objective data. The objective of this project is to evaluate, by mean of oropharyngoesophageal scintigraphy (OPES), the impact of an occluded tracheal tube on swallowing of patients treated for head and neck cancer before hospital discharge, to provide further knowledges especially useful for the out-patient care management.

The present study was designed as a cross-sectional observational study providing the enrollment of tracheostomized patients undergoing major oncological surgery for head-neck cancer.

ELIGIBILITY:
Inclusion criteria

* Age >18 years
* Tracheal tube diameter of 5.0 mm and outside diameter of 9.4 mm
* Tolerance of the tracheal tube capping for almost 48 hours without pathologic desaturation during continue monitoring of SpO2
* Ability to swallow in accordance to the inpatient training program
* Ability to suck with a straw without oral leakage Exclusion criteria
* Previous head and neck radiotherapy
* Patients with nasal tube feeding
* Patients with poor cognition or poor general condition or affected by neurological o other nontumor-related dysphagia
* Patients total laryngectomized
* Patients unable to maintain the orthostatic position

Ages: 18 Years to 70 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: In this study, a total of 20 tracheostomized patients undergoing primary major surgery for head and neck cancer will be enrolled at the Otolaryngology hospitalization department of the Fondazione Policlinico Univesitario A. Gemelli, in Rome (Italy)
Sampling Method: Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2021-12-06 (Actual); Primary Completion 2026-10-06 (Estimated); Study Completion 2026-10-06 (Estimated)

PRIMARY OUTCOMES:
To provide objective data on the bolus transit during swallowing in tracheostomized patients with tracheal tube and without tracheal tube | five years
  To provide objective data on the bolus transit during swallowing in tracheostomized patients with tracheal tube and without tracheal tube closing directly the tracheal stoma with a plaster, in order to sustain the choice to preserve the TT in dysphagic patients after oncologic surgery for more security during swallowing rehabilitation or adjuvant treatment.

SECONDARY OUTCOMES:
To evaluate the features of swallowing | five years
  To evaluate the features of swallowing, specifically bolus transit, in patients affected by head and neck cancer who underwent major oncological surgery.

CONTACTS AND LOCATIONS:
Overall Officials: Jacopo Galli, Principal Investigator — Fondazione Policlinico Universitario A. Gemelli IRCCS - Roma
Locations (1):
- Maria Raffaella Marchese, Roma, Italy

IPD SHARING:
Plan to Share IPD: No